CLINICAL TRIAL: NCT02779933
Title: Epidemiology of Risk Factors for Hospital-acquired Pneumonia in ICU Patients
Brief Title: Epidemiology of Risk Factors for Hospital-acquired Pneumonia (HAP) in Intensive Care Unit (ICU) Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Radovan Uvizl, MUDr., Ph.D., University Hospital Olomouc
Other Study IDs: 63/16
Record Dates: First submitted 2016-05-12; First posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Hospital-acquired Pneumonia; Epidemiology; Risk Factors
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — endotracheal aspirate
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Epidemiology od HAP — no intervention

SUMMARY:
A retrospective, observational study compiled data from all consecutively admitted patients older than 18 years at ICU University Hospital in Olomouc in the period from 1 January 2011 to 31 December 2015 who fulfilled the criteria of HAP. The aim was to determine the severity of the specific risk factors of early and late HAP. Risk factors were divided into factors from the patient and from the hospitalization. Furthermore, an assessment of their relationship to mortality.

DETAILED DESCRIPTION:
The primary outcome was to evaluate the relationship between risk factors and the development of early/late onset HAP. Another outcome was assessed to evaluate the relation of risk factors early/late onset HAP and mortality. The crucial time for evaluating the presence of risk factors was their presence from hospital admission to the moment of fulfilling the criteria for pneumonia. Risk factors were divided into two groups, on factors of the patient (uncontrollable) and by the hospitalization (controllable). Factors of the patient were: gender (male/female), age at enrollment (years), Acute Physiology and Chronic Health Evaluation II (APACHE II) score, multi-organ failure presence (MOF), hypertension, ischemic heart disease (IHD) chronic renal insufficiency (CRI), continual use of renal replacement therapy (CRRT), acute renal insufficiency (ARI), diabetes mellitus (DM), Chronical Obstructive Pulmonary Disease (COPD), immunosuppression or leukopenia <1.5x109/l, impaired consciousness with Glasgow coma scale (GCS) <8 tracheotomy, head trauma/neurosurgery, abdominal surgery-thoracotomy. Side factors hospitalization were: aspiration into the lungs, urgent intubation, reintubated, sedation, bronchoscopy, nasogastric intubation, enteral feeding continuously/intermittently intolerance of enteral nutrition, physiotherapy, repeated transport of the patient from the ICU, length of hospital stay, length of mechanical ventilation, 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Hospital-Acquired Pneumonia
* Intensive Care patient
* X-ray signs of pneumonia

Exclusion Criteria:

* Age less than 18 years
* Negative culture findings in the airways
* Low quantity of culture findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients hospitalized in the ICU Department of Anesthesiology and Intensive Care Medicine, UH Olomouc. On inclusion did not affect the method of ensuring lower airways (invasive/non-invasive) or results (positivity/negativity) taken microbiological samples from the lower airways (endobronchial aspirate or bronchoalveolar lavage) as approximately one third of samples can be microbiologically negative even when overt bronchopneumonia. Patient cohort consisted of all patients older than 18 years who met the clinical criteria and HAP were consecutively admitted to the ICU.
Sampling Method: Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
30-day mortality (non modifiable HAP risk factor) | 30 days
  Yes/No assessment

SECONDARY OUTCOMES:
Duration of mechanical ventilation before onset of HAP (non modifiable HAP risk factor) | 7 days
  Assessment if mechanical ventilation was provided, or for how long
Duration of hospital stay before onset of HAP (non modifiable HAP risk factor) | 7 days
  Assessment if hospital stay was present, or for how long
Repeated transport of the patient from the ICU (non modifiable HAP risk factor) | 30 days
  Assessment if repeated transports were present or not
Implementation of physiotherapy before onset of HAP (non modifiable HAP risk factor) | 7 days
  Assessment if physiotherapy was provided or not
Intolerance of enteral nutrition before onset of HAP (non modifiable HAP risk factor) | 7 days
  Yes/No assessment
Nasogastric intubation before onset of HAP (non modifiable HAP risk factor) | 7 days
  Yes/No assessment
Bronchoscopy before onset of HAP (non modifiable HAP risk factor) | 7 days
  Yes/No assessment
Sedation administration before onset of HAP (non modifiable HAP risk factor) | 7 days
  Yes/No assessment
Urgent tracheal intubation before onset of HAP (non modifiable HAP risk factor) | 7 days
  Yes/No assessment
Tracheal reintubation before onset of HAP (non modifiable HAP risk factor) | 7 days
  Yes/No assessment
Aspiration into the lungs before onset of HAP (non modifiable HAP risk factor) | 7 days
  Yes/No assessment
Condition after abdominal surgery or thoracotomy before onset of HAP (modifiable HAP risk factor) | 7 days
Condition after head trauma or neurosurgery before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Condition after tracheotomy before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Impaired consciousness with Glasgow coma scale low than 8 before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Immunosuppression or leukopenia less than 1.5x10 9/L before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Chronical Obstructive Pulmonary Disease before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Diabetes mellitus before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Acute renal insufficiency without renal replacement therapy before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Acute renal insufficiency with renal replacement therapy before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Chronic renal insufficiency before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Ischemic heart disease before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Hypertension before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment
Multi-organ failure before onset of HAP (modifiable HAP risk factor) | 7 days
  Yes/No assessment

CONTACTS AND LOCATIONS:
Overall Officials: Radovan Uvizl, Principal Investigator — UH Olomouc, Czech Republic

IPD SHARING:
Plan to Share IPD: Yes
Collecting data from individual patients medical documentation

REFERENCES:
- [Derived] Uvizl R, Kolar M, Herkel T, Vobrova M, Langova K. Possibilities for modifying risk factors for the development of hospital-acquired pneumonia in intensive care patients: results of a retrospective, observational study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2017 Sep;161(3):303-309. doi: 10.5507/bp.2017.019. Epub 2017 Apr 26. PMID 28461706